CLINICAL TRIAL: NCT04119622
Title: A Phase II Study of XELOX and Toripalimab in the Neoadjuvant Treatment of Stage II/III Gastric or GE Junction Adenocarcinoma
Brief Title: Toripalimab Combined With Chemotherapy as Neoadjuvant Treatment of Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO63
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Gastric Cancer Stage II; Gastric Cancer Stage III
Keywords: Toripalimab; JS001; Gastric Cancer; neoadjvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — toripalimab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- XELOX combined with Toripalimab (Experimental)
  Interventions: Drug: Toripalimab; Drug: oxaliplatin; Drug: capecitabine

INTERVENTIONS:
Drug: Toripalimab — toripalimab 240 mg d1; q3w, up to two cycles.
Drug: oxaliplatin — oxaliplatin 130 mg/m2 QD, d1,q3w, up to two cycles
Drug: capecitabine — apecitabine 1000 mg/m2 BID, d1-d14 ,q3w, up to two cycles

SUMMARY:
Gastric cancer (GC) is one of the most common malignancies. According to the global cancer statistics 2018, there were 1,033,701 new cases of gastric cancer per year, ranked the fifth place in new tumors, and 782,685 deaths, ranked the second place in cancer deaths. At present, surgery is the only way to cure gastric cancer, but the 5-year survival rate is only 20%-30%. studies have confirmed that neoadjuvant therapy could improve the R0 resection rate and overall survival, which is considered a better treatment strategy.

PD 1 monoclonal antibody is definitely effective in neoadjuvant therapy in other tumors such as NSCLC and bladder cancer, especially in PD-L1+ patients. However, there is no research of PD-1 monoclonal antibody in neoadjuvant therapy of gastric cancer. Thus we plan to conduct this prospective phase II clinical trial, evaluating the safety and efficacy of toripalimab, also known as JS001, in combination with XELOX for the neoadjuvant therapy of gastric cancer.

DETAILED DESCRIPTION:
This phase II trial is a single-arm, open Label, non-randomized and single-center clinical study. Patients who met the study criteria will receive the combination of toripalimab (240 mg d1) with XELOX (oxaliplatin 130 mg/m2 QD, d1, capecitabine 1000 mg/m2 BID, d1-d14) of a 3-week treatment cycle up to two cycles. After the second cycle of treatment, clinical efficacy evaluation will be done by MDT according to iRECIST. For patients with CR/PR/SD, surgery will be performed within 4 weeks. For patients with disease progress, MDT will determine whether the surgery could be performed. If resection could not be done, the patients would receive Original chemotherapy with toripalimab for 1 more cycle, chemoradiotherapy or the second line chemotherapy. The primary endpoint is Major pathological response.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma, siwert type I was excluded.
2. Clinical determined T3/4 N any or T 1/2 N 2/3 referred to AJCC 8, based on CT, gastroscopy, endoscopic ultrasound, gastrointestinal angiography, general ultrasound, or laparoscope if the patient can afford.
3. No prior chemotherapy and/or immunotherapy and/or radiation therapy.
4. Age 18 to 75 years old.
5. ECOG 0 or 1 .
6. Adequate Organ Function Laboratory Values Hb≥90g/L, WBC≥3.5×109 /L, ANC≥1.5×109 /L, Platelets≥100×109 /L Serum creatinine ≤1.0×ULN ALT≤1.5 ×UNL , AST ≤1.5×ULN，ALP≤ 1.5 ×ULN Serum total bilirubin ≤1.5 × ULN
7. Signed Informed consent

Exclusion Criteria:

1. Pathology types other than adenocarcinoma, such as squamous cell carcinoma.
2. intra-abdominal dissemination or distant metastasis (M1).
3. Digestive tract obstruction or repeated bleeding which can not be controlled, clinically significant ascites.
4. Those who cannot swallow pills.
5. Cirrhosis caused by any cause.
6. Heart function NYHA > I degree
7. Previous myocardial infarction, unstable angina, stroke and uncontrolled arrhythmia.
8. with any contraindications for surgery.
9. Previously received chemotherapy and or radiation therapy.
10. Previously received any anti-PD 1 , anti - PD L1/L2 antibodies, anti-CTLA 4 antibodies and other immunotherapy.
11. Previously received other anti-tumor treatments.
12. History of surgical resection for gastric cancer.
13. Have had other tumors in the past, except for cured skin cancer and cervical cancer in situ.
14. Accompanied by systemic diseases which cannot meet the conditions of chemotherapy.
15. Pregnancy and lactating patients.
16. History of mental diseases.
17. Poor compliance.
18. Active central nervous system (CNS) metastases and/or carcinomatous meningitis.
19. History of gastrointestinal perforation and/or fistula in the past 6 months; history of intestinal obstruction (including incomplete intestinal obstruction which need for extraintestinal Nutritional); inflammatory bowel disease or extensive bowel resection(Partial colon resection or extensive small Intestinal resection complicated with chronic diarrhea);Crohn's disease; ulcerative colitis or chronic diarrhea.
20. History of interstitial pneumonia, drug-induced pneumonia, idiopathic pneumonia or active pneumonia.
21. Active tuberculosis (TB), undergoing anti-tuberculosis treatment or within 1 year before the first dose
22. has infected Human immunodeficiency virus (HIV1 / 2 antibody positive).
23. Has known active hepatitis B or hepatitis C. Acute or chronic active hepatitis B or hepatitis C virus infection, hepatitis B virus (HBV) DNA > 2000 IU / ml or 10^4 copies / ml; Hepatitis C virus (HCV) RNA > 10^3 copies / ml ; hepatitis B surface antigen(HbsAg) and anti-HCV antibody is positive at the same time.
24. Severe infections active or poorly controlled. Severe infections within 4 weeks before the first dose, includes but not limited to hospitalization attributed to infection, bacteremia or severe pneumonia complications.
25. Active autoimmune disease requiring systemic treatment or the history within 2 years (one with vitiligo, psoriasis, alopecia or Graves' disease not requiring systemic treatment in the last 2 years, hypothyroidism only requiring thyroid hormones alternative treatment and type 1 diabetes only requiring insulin replacement therapy can be enrolled). Have has known history of primary immunodeficiency. patients with positive autoimmune antibodies only will need to be confirmed the presence of autoimmune diseases according to the investigator's judgment.
26. Application of immunosuppressive drugs within the latest 4 weeks, excluding nasal glucocorticoids and topical glucocorticoids by inhaling or other routings. Physiological doses of systemic glucocorticoids (prednisone not exceeding 10 mg/day or equivalent dose of other glucocorticoids) and temporary use of glucocorticoids for the treatment of dyspnea caused by asthma, chronic obstructive pulmonary disease and other diseases would be allowed.
27. have received live attenuated vaccines within 4 weeks or intend to be vaccinated during the study period.
28. have received systemic immunostimulant treatment within 4 weeks.
29. Have undergone major surgery (such as craniotomy, thoracotomy or laparotomy) within 4 weeks, or unhealed wound, ulcer or fracture at present.
30. Have uncontrolled metabolic disorders , other non-malignant tumors, systemic diseases or secondary reactions originated from the cancer which may lead to higher medical risks and/or the uncertainty of survival evaluation.
31. patients with other acute or chronic diseases, psychiatric disorders, or abnormal laboratory tests that may lead to the increasing risk of participating the research and drug administration, or interference results Interpretation, whom may be excluded from the study according to the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate | Up to 6 months
  Proportion of subjects with residual tumor less than 10% or complete response

SECONDARY OUTCOMES:
Incicende of Adverse Events (AEs) | Up to 6 months
  Number of patients with AE, treatment-related AE (TRAE), immune-related AEs (irAE), AE of special interest (AESI), serious adverse event (SAE) assessed by CTCAE v5.0.
Pathologic Complete Response (pCR) Rate | Up to 6 months
  Proportion of subjects with absence of viable tumor on surgical resection specimen as determined by local pathology review.
Overall Response Rate (ORR) | Up to 6 months
  Proportion of subjects with initial RECIST 1.1 measurable disease who have complete response (CR) or partial response (PR) according to iRECIST
Disease Free Survival (DFS) | Up to 5 years
  Time from Cycle 1 Day 1 treatment administration to the first documented event of: disease progression, disease recurrence following surgery (preferably biopsy proven), or death - whichever occurs first.
Overall Survival (OS) | Up to 5 years
  Time from Cycle 1 Day 1 treatment administration to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences, Beijing